CLINICAL TRIAL: NCT00117559
Title: Improving Quality of Life for Veterans Undergoing Interferon Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F3332-P
Record Dates: First submitted 2005-06-30; First posted 2005-07-07 (Estimated); Results first posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Depression; Hepatitis C
Keywords: Psychotherapy,group; Rehabilitation; Telecommunications
MeSH Terms: conditions — Depression; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TEL-CBT (Experimental): Telehealth, problem solving based treatment provided over the telephone
  Interventions: Behavioral: Telehealth Treatment
- Treatment as Ususal (No Intervention): Control group, no treatment provided

INTERVENTIONS:
Behavioral: Telehealth Treatment — Participants receive a 15-minute telephone call for 8 weeks
  Arms: TEL-CBT

SUMMARY:
The purpose of this study is to evaluate a group psychotherapy intervention and a telehealth intervention for veterans undergoing interferon treatment for the hepatitis C virus. It is hypothesized that the cognitive behavioral therapy (CBT) condition and the telehealth condition will result in significantly improved outcomes, including enhanced adherence, quality of life, and psychological status.

DETAILED DESCRIPTION:
The purpose of the proposed pilot study is to evaluate a rehabilitative cognitive-behavioral group psychotherapy intervention and a telehealth intervention for veterans undergoing interferon treatment for the hepatitis C virus (HCV). The specific objectives of the proposed pilot study are: 1) develop study methods and materials; 2) evaluate study feasibility; and 3) assess the efficacy of a cognitive-behavioral group therapy approach and a telehealth approach as compared to care as usual in a randomized design. Participants will be 45 patients (15 participants in each condition) from the VA Boston Healthcare System who are undergoing interferon treatment for HCV. Assessment will occur at pre-treatment, post-treatment, and 3-month follow-up. Assessments will measure key areas, including adherence, quality of life, and psychological distress. Analyses will examine study feasibility and the effects of the treatment condition. It is hypothesized that the CBT condition and the telehealth condition will result in significantly improved outcomes, including enhanced adherence, quality of life, and psychological status. This treatment approach addresses initiatives by the National VHA Hepatitis C Program by optimizing the care of veterans experiencing the devastating side effects of interferon treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hepatitis C.
* Must be on the interferon treatment
* Need to have access to telephone.

Exclusion Criteria:

* Life threatening or acute illness
* Current alcohol or substance abuse or dependence
* Individuals already receiving psychological interventions specifically to manage the side effects of the IFN treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Silberbogen, PhD, Principal Investigator — VA Medical Center, Jamaica Plain Campus
Locations (1):
- VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TEL-CBT: Telehealth, problem solving based treatment
  Telehealth Treatment: Participants receive a 15-minute telephone call for 8 weeks
- Treatment as Usual: Control group
Period: Overall Study
Arm/Group | TEL-CBT | Treatment as Usual
Started | 9 | 10
Completed | 8 | 9
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEL-CBT | Treatment as Usual | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.78 (4.35) | 54.50 (6.38) | 54.16 (5.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
BDI [Mean (Standard Deviation); unit: units on a scale] | 12.93 (8.17) | 12.29 (10.10) | 12.61 (9.14)

OUTCOME MEASURES:

1. Primary Outcome: BDI
Description: Beck Depression Inventory - measures depression. Range for Total score = 0 to 63 Higher scores are indicative of increased depression
  The Beck Depression Inventory (BDI; Beck & Steer, 1988) is a widely used 21-item self-report instrument designed to assess depressive mood and symptoms. Each item is rated on a 4-point scale ranging from 0 to 3, with higher scores reflecting greater severity of depressive symptoms for the past two weeks. A sample item is "I do not feel sad." The BDI has demonstrated reliability (split-half reliability coefficient of .93) and validity (correlations with clinician ratings of depression range from .62 to .75; Beck, Steer, & Garbing, 1988). Cronbach's alpha was high for the present sample at both time points (a = .91 and .90).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TEL-CBT | Treatment as Usual
Number analyzed (Participants) | 8 | 9
units on a scale
  Pre-Treatment | 12.93 (8.17) | 12.29 (10.10)
  Post-Treatment | 10.45 (6.03) | 16.67 (9.80)
Statistical Analysis 1: Comparison: TEL-CBT vs Treatment as Usual; Test type: Superiority or Other; p < .05, ANOVA

ADVERSE EVENTS:
Time Frame: During recruitment and when running subjects
Groups:
- Treatment as Ususal: Control group
Arm/Group | TEL-CBT | Treatment as Ususal
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 0/10

LIMITATIONS AND CAVEATS:
Small sample size, all male, no in-person comparison group, reporting bias in self-report measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No